CLINICAL TRIAL: NCT02135640
Title: A Randomized, Single-blind, Parallel-group, Placebo-controlled, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Denosumab Administered Subcutaneously to Healthy Adults in China
Brief Title: China HVT Safety, PK, PD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114197
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- denosumab 60 mg (Experimental): solution
  Interventions: Drug: denosumab 60mg
- denosumab 120 mg (Experimental): solution
  Interventions: Drug: denosumab 120 mg
- placebo (Placebo Comparator): solution
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: denosumab 60mg — solution
  Arms: denosumab 60 mg
Drug: denosumab 120 mg — solution
  Arms: denosumab 120 mg
Drug: placebo — solution
  Arms: placebo

SUMMARY:
This study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of denosumab administered subcutaneously to healthy adults in China.

DETAILED DESCRIPTION:
Denosumab is a fully human monoclonal IgG2 antibody to RANKL that being investigated as a therapeutic agent in all bone diseases characterized by excessive bone resorption, such as primary and secondary osteoporosis, metastatic bone diseases, and other diseases involving bone loss associated with increases in osteoclast function. This will be a single-blind, placebo-controlled single-dose study. All subjects will be randomized to denosuamb 60 mg, denosumab 120 mg or placebo in a ration of 3:3:2. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of denosumab administered subcutaneously to healthy adults in China. The primary endpoints for safety are: subject incidence of treatment-emergent adverse events, including clinically significant changes in physical examinations, laboratory safety tests, ECG and vital signs. The secondary endpoints are PK and PD (s-CTX1) parameter estimates.

ELIGIBILITY:
Inclusion Criteria:

* Resident in China and of Chinese ancestry.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin > 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age, inclusive, from date of birth, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. In questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (< 140 pmol/L) is confirmatory.

OR Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for the duration of the study and for a minimum of 6 months after the last dose of study medication.

* Body weight of at least 50 kg and body mass index (BMI) from 19 to 24 kg/m2 at time of screening.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A prior history or current evidence of osteomyelitis or ONJ.
* An active dental or jaw condition that requires oral surgery.
* A planned invasive dental procedure during the course of the study.
* A non-healed dental or oral surgery.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* A positive test for syphilis at Screening.
* Abnormal serum calcium: current hypocalcemia or hypercalcemia. Albumin-adjusted serum calcium levels must be within the normal range of the central laboratory.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of > 14 drinks/week for men or > 7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 150 ml (5 ounces) of table wine or 360 ml (12 ounces) of beer or 45 ml (1.5 ounces) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, especially known sensitivity to mammalian-derived drug preparations, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum human chorionic gonadotropin (hCG) test at screening or urine hCG test prior to dosing (day -1).
* A chest X-ray or computed tomography (CT) scan that reveals evidence of clinical significant abnormalities e.g., tuberculosis. A chest X-ray must be taken at Day-1 if a chest X-ray or CT scan is not available within 6 months prior to that day.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Significant changes in physical activity during the 6 months before study drug administration or constant levels of intense physical exercise.
* Prior use of medications within 4 weeks or 5 half-lives (whichever period is greater) before and during the study. This includes medications such as, but not limited to:

Estrogen-containing contraceptives Bisphosphonates Fluoride Hormone replacement therapy (i.e., tibolone, estrogen, estrogen-like compounds such as raloxifene) Calcitonin Strontium Parathyroid hormone or derivatives Supplemental vitamin D (>1000 IU/day) Glucocorticosteroids (inhaled or topical corticosteroids administered more than 2 weeks prior to enrolment are allowed) Anabolic steroids Calcitriol Diuretics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07-17 (Actual); Primary Completion 2015-02-17 (Actual); Study Completion 2015-02-17 (Actual)

PRIMARY OUTCOMES:
adverse events | up to 26 weeks
  subjects incidence of treatment adverse events, including clinically-significant changes in physical examinations, laboratory safety tests, ECG and vital signs

SECONDARY OUTCOMES:
PK parameter estimates | up to 19 weeks
  Cmax, Tmax, AUC(0-t),
PD parameter estimateds | up to 19 weeks
  serum CTX1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

REFERENCES:
- [Derived] Chen Q, Hu C, Liu Y, Song R, Zhu W, Zhao H, Nino A, Zhang F, Liu Y. Pharmacokinetics, pharmacodynamics, safety, and tolerability of single-dose denosumab in healthy Chinese volunteers: A randomized, single-blind, placebo-controlled study. PLoS One. 2018 Jun 22;13(6):e0197984. doi: 10.1371/journal.pone.0197984. eCollection 2018. PMID 29933364
- See also: Results for study 114197 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114197?search=study&study_ids=114197#rs